CLINICAL TRIAL: NCT00060320
Title: A Phase III Double-Blind, Randomized, Placebo-Controlled Crossover Trial Of Black Cohosh In The Management Of Hot Flashes
Brief Title: Black Cohosh in Treating Hot Flashes in Women Who Have or Who Are At Risk of Developing Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: NCCTG-N01CC; CDR0000301615 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-05-06; First posted 2003-05-07 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer; Hot Flashes
Keywords: stage IV breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; hot flashes
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes | interventions — black cohosh root extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- black cohost (Experimental): Patients receive oral black cohosh twice daily for 4 weeks. All patients then cross over to the other arm and receive treatment for 4 weeks.
  After completion of the crossover treatment, all patients may opt to receive open-label black cohosh for an additional 8 weeks.
  Patients complete a hot flash diary daily at baseline and during the 8-week double-blind study, and then daily for 8 weeks during optional open-label treatment.
  Patients who opt to receive open-label black cohosh are followed at 6 months, 1 year, and 2 years.
  Interventions: Dietary Supplement: black cohosh; Other: placebo
- placebo (Placebo Comparator): Patients receive oral placebo twice daily for 4 weeks. All patients then cross over to the other arm and receive treatment for 4 weeks.
  After completion of the crossover treatment, all patients may opt to receive open-label black cohosh for an additional 8 weeks.
  Patients complete a hot flash diary daily at baseline and during the 8-week double-blind study, and then daily for 8 weeks during optional open-label treatment.
  Patients who opt to receive open-label black cohosh are followed at 6 months, 1 year, and 2 years.
  Interventions: Dietary Supplement: black cohosh; Other: placebo

INTERVENTIONS:
Dietary Supplement: black cohosh
Other: placebo

SUMMARY:
RATIONALE: The herbal supplement black cohosh may be effective in relieving hot flashes in women.

PURPOSE: Randomized phase III trial to determine the effectiveness of black cohosh in relieving hot flashes in women who have breast cancer or who are at risk of developing breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of black cohosh vs placebo in diminishing hot flash activity in women with breast cancer OR a concern about taking hormones because of a fear of breast cancer.
* Determine whether continued use of this drug by these patients leads to prolonged reduction of the hot flash score with minimal toxic effects.
* Correlate the reduction of hot flash score with improvement in quality of life and related outcomes in patients treated with this drug.
* Determine the toxic effects of this drug in these patients.
* Determine whether abnormal sweating is decreased in patients treated with this drug.

OUTLINE: This is a randomized, double-blind, placebo-controlled, crossover study. Patients are stratified according to age (18 to 49 vs 50 and over), current tamoxifen use (yes vs no vs unknown), current raloxifene use (yes vs no vs unknown), current aromatase inhibitor use (yes vs no), duration of hot flash symptoms (less than 9 months vs 9 months or more), and average frequency of hot flashes per day (2-3 vs 4-9 vs 10 or more). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral black cohosh twice daily for 4 weeks.
* Arm II: Patients receive oral placebo twice daily for 4 weeks. All patients then cross over to the other arm and receive treatment as above for 4 weeks.

After completion of the crossover treatment, all patients may opt to receive open-label black cohosh for an additional 8 weeks.

Patients complete a hot flash diary daily at baseline and during the 8-week double-blind study, and then daily for 8 weeks during optional open-label treatment.

Patients who opt to receive open-label black cohosh are followed at 6 months, 1 year, and 2 years.

PROJECTED ACCRUAL: A total of 110 patients (55 patients per arm) will be accrued for this study within 6-11 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* History of breast cancer OR concern about taking hormones because of fear of breast cancer

  * No current active disease
  * No current evidence of malignant disease
* Bothersome hot flashes

  * Patient-reported occurrence at least 14 times per week and of sufficient severity to make the patient desire therapeutic intervention
* Hormone receptor status:

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Performance status

* ECOG 0-1

Life expectancy

* At least 6 months

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to complete questionnaires alone or with assistance

PRIOR CONCURRENT THERAPY:

Chemotherapy

* More than 4 weeks since prior antineoplastic chemotherapy
* No concurrent antineoplastic chemotherapy during the double-blind portion of the study

Endocrine therapy

* More than 4 weeks since prior androgens, estrogens, or progestational agents
* More than 2 weeks since prior dehydroepiandrosterone (DHEA) for hot flashes
* No concurrent androgens, estrogens, or progestational agents during the double-blind portion of the study
* No concurrent DHEA for hot flashes
* Concurrent tamoxifen, raloxifene, or an aromatase inhibitor is allowed provided the patient started the drug at least 4 weeks prior to study entry and plans to continue the drug throughout the double-blind portion of the study Other
* More than 2 weeks since prior antidepressants
* More than 2 weeks since other prior agents for treating hot flashes (e.g., clonidine or Bellergal-s)
* No prior black cohosh
* No concurrent antidepressants during the double-blind portion of the study
* No other concurrent agents for treating hot flashes (e.g., clonidine or Bellergal-s)

  * Concurrent vitamin E and/or soy allowed provided patient is on a stable dose for at least 1 month prior to study entry and plans to continue the same dose throughout study duration
* No concurrent oral herbal therapies or therapeutic herbal teas or tinctures except beverage teas (e.g., chamomile, ginger, peppermint, lemongrass, and fruit-based tea)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2003-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Hot flash activity | Up to 3.5 years

SECONDARY OUTCOMES:
Reduction of hot flash score | Up to 3.5 years
Quality of life | Up to 3.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Barbara A. Pockaj, MD, Study Chair — Mayo Clinic Hospital
Locations (13):
- United States (13):
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Result] Pockaj BA, Gallagher JG, Loprinzi CL, Stella PJ, Barton DL, Sloan JA, Lavasseur BI, Rao RM, Fitch TR, Rowland KM, Novotny PJ, Flynn PJ, Richelson E, Fauq AH. Phase III double-blind, randomized, placebo-controlled crossover trial of black cohosh in the management of hot flashes: NCCTG Trial N01CC1. J Clin Oncol. 2006 Jun 20;24(18):2836-41. doi: 10.1200/JCO.2005.05.4296. PMID 16782922